CLINICAL TRIAL: NCT00003322
Title: A Phase III Randomized Trial of Intravenous Paclitaxel and Cisplatin Versus Intravenous Paclitaxel, Intraperitoneal Cisplatin and Intraperitoneal Paclitaxel in Patients With Optimal Stage III Epithelial Ovarian Carcinoma or Primary Peritoneal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Primary Peritoneal or Stage III Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066273; GOG-0172
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells. It is not yet known whether intravenous two-drug combination chemotherapy is more effective than intravenous and intraperitoneal infusions of three-drug combination chemotherapy for treating primary peritoneal or stage III epithelial ovarian cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of intravenous two-drug combination chemotherapy with intravenous and intraperitoneal three-drug combination chemotherapy in treating patients who have primary peritoneal or stage III epithelial ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare pathological response, recurrence-free interval, and survival in patients with optimal stage III epithelial ovarian cancer or primary peritoneal carcinoma receiving intravenous (IV) paclitaxel and cisplatin vs IV paclitaxel and intraperitoneal (IP) cisplatin plus IP paclitaxel. II. Compare the toxic effects and complications of these 2 treatment regimens in these patients. III. Determine the frequency and prognostic significance of BRCA1 and BRCA2 mutations in these patients. IV. Determine the effect of non-genetic risk factors on the course of disease in BRCA1- and BRCA2-related ovarian cancer or primary peritoneal carcinoma. V. Compare the quality of life of these patients receiving these treatments.

OUTLINE: This is a randomized study. Patients are stratified according to gross residual disease (present vs absent) and whether second-look surgery will be performed at the end of treatment (yes vs no). Blood is drawn for BRCA mutation analysis and DNA extraction before the start of chemotherapy, but after randomization. Patients are randomized to one of two treatment arms. Patients in arm I receive IV paclitaxel by 24-hour infusion on day 1 followed by IV cisplatin on day 2. Patients in arm II receive IV paclitaxel by 24-hour infusion on day 1 followed by intraperitoneal (IP) cisplatin on day 2, plus IP paclitaxel on day 8. Treatment for both arms repeats every 3 weeks for a total of 6 treatment courses. Following chemotherapy, second look surgery is performed if selected by the patient. Quality-of-life assessments are performed prior to randomization, prior to course 4, 3-6 weeks after the completion of course 6 and prior to second look surgery if selected, 6 months after treatment is completed, and 12 months after treatment is completed. Patients are followed every 3 months for 2 years, then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 384 patients will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven primary peritoneal carcinoma or optimal (no greater than 1 cm residual disease) stage III epithelial ovarian carcinoma with the following epithelial cell types: Serous adenocarcinoma Endometrioid adenocarcinoma Mucinous adenocarcinoma Undifferentiated carcinoma Clear cell adenocarcinoma Mixed epithelial carcinoma Transitional cell carcinoma Malignant Brenner's Tumor Adenocarcinoma NOS Prior surgery for ovarian/peritoneal carcinoma required No epithelial ovarian carcinoma of low malignant potential (borderline carcinoma)

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal No acute hepatitis Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No unstable angina No myocardial infarction within prior 6 months Patients with abnormal cardiac conduction are eligible if disease stable for at least 6 months Other: No septicemia or severe infection No severe gastrointestinal bleeding No other invasive malignancy within past 5 years except nonmelanoma skin cancer Any previous cancer treatment must not contraindicate this protocol therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics No more than 6 weeks since prior surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 1998-03; Primary Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah K. Armstrong, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (67):
- United States (66):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Barlin JN, Dao F, Bou Zgheib N, Ferguson SE, Sabbatini PJ, Hensley ML, Bell-McGuinn KM, Konner J, Tew WP, Aghajanian C, Chi DS. Progression-free and overall survival of a modified outpatient regimen of primary intravenous/intraperitoneal paclitaxel and intraperitoneal cisplatin in ovarian, fallopian tube, and primary peritoneal cancer. Gynecol Oncol. 2012 Jun;125(3):621-4. doi: 10.1016/j.ygyno.2012.03.027. Epub 2012 Mar 21. PMID 22446622
- [Background] Rubatt JM, Darcy KM, Tian C, Muggia F, Dhir R, Armstrong DK, Bookman MA, Niedernhofer LJ, Deloia J, Birrer M, Krivak TC. Pre-treatment tumor expression of ERCC1 in women with advanced stage epithelial ovarian cancer is not predictive of clinical outcomes: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 May;125(2):421-6. doi: 10.1016/j.ygyno.2012.01.008. Epub 2012 Jan 16. PMID 22261301
- [Background] Tian C, Ambrosone CB, Darcy KM, Krivak TC, Armstrong DK, Bookman MA, Davis W, Zhao H, Moysich K, Gallion H, DeLoia JA. Common variants in ABCB1, ABCC2 and ABCG2 genes and clinical outcomes among women with advanced stage ovarian cancer treated with platinum and taxane-based chemotherapy: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 Mar;124(3):575-81. doi: 10.1016/j.ygyno.2011.11.022. Epub 2011 Nov 21. PMID 22112610
- [Background] Hamilton CA, Miller A, Miller C, Krivak TC, Farley JH, Chernofsky MR, Stany MP, Rose GS, Markman M, Ozols RF, Armstrong DK, Maxwell GL. The impact of disease distribution on survival in patients with stage III epithelial ovarian cancer cytoreduced to microscopic residual: a Gynecologic Oncology Group study. Gynecol Oncol. 2011 Sep;122(3):521-6. doi: 10.1016/j.ygyno.2011.04.041. Epub 2011 Jun 17. PMID 21683993
- [Background] Aletti GD, Nordquist D, Hartmann L, Gallenberg M, Long HJ, Cliby WA. From randomized trial to practice: single institution experience using the GOG 172 i.p. chemotherapy regimen for ovarian cancer. Ann Oncol. 2010 Sep;21(9):1772-1778. doi: 10.1093/annonc/mdq025. Epub 2010 Feb 5. PMID 20139154
- [Background] von Gruenigen VE, Huang HQ, Gil KM, Gibbons HE, Monk BJ, Rose PG, Armstrong DK, Cella D, Wenzel L. A comparison of quality-of-life domains and clinical factors in ovarian cancer patients: a Gynecologic Oncology Group study. J Pain Symptom Manage. 2010 May;39(5):839-46. doi: 10.1016/j.jpainsymman.2009.09.022. PMID 20471545
- [Background] Darcy KM, Tian C, Ambrosone CB, et al.: A Gynecologic Oncology Group study of associations between polymorphisms in ABC transporter genes (ABCB1, ABCC2, and ABCG2) and outcome in advanced stage epithelial ovarian cancer treated with platinum and taxane chemotherapy. [Abstract] J Clin Oncol 27 (Suppl 15): A-5567, 2009.
- [Background] Farley JH, Tian C, Rose GS, Brown CL, Birrer M, Maxwell GL. Race does not impact outcome for advanced ovarian cancer patients treated with cisplatin/paclitaxel: an analysis of Gynecologic Oncology Group trials. Cancer. 2009 Sep 15;115(18):4210-7. doi: 10.1002/cncr.24482. PMID 19536873
- [Background] Zorn KK, Tian C, McGuire WP, Hoskins WJ, Markman M, Muggia FM, Rose PG, Ozols RF, Spriggs D, Armstrong DK. The prognostic value of pretreatment CA 125 in patients with advanced ovarian carcinoma: a Gynecologic Oncology Group study. Cancer. 2009 Mar 1;115(5):1028-35. doi: 10.1002/cncr.24084. PMID 19156927
- [Background] Havrilesky LJ, Secord AA, Darcy KM, Armstrong DK, Kulasingam S; Gynecologic Oncology Group. Cost effectiveness of intraperitoneal compared with intravenous chemotherapy for women with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2008 Sep 1;26(25):4144-50. doi: 10.1200/JCO.2007.13.1961. PMID 18757328
- [Background] Bristow RE, Santillan A, Salani R, Diaz-Montes TP, Giuntoli RL 2nd, Meisner BC, Armstrong DK, Frick KD. Intraperitoneal cisplatin and paclitaxel versus intravenous carboplatin and paclitaxel chemotherapy for Stage III ovarian cancer: a cost-effectiveness analysis. Gynecol Oncol. 2007 Sep;106(3):476-81. doi: 10.1016/j.ygyno.2007.05.043. Epub 2007 Aug 3. PMID 17688927
- [Background] Winter WE 3rd, Maxwell GL, Tian C, Carlson JW, Ozols RF, Rose PG, Markman M, Armstrong DK, Muggia F, McGuire WP; Gynecologic Oncology Group Study. Prognostic factors for stage III epithelial ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Aug 20;25(24):3621-7. doi: 10.1200/JCO.2006.10.2517. PMID 17704411
- [Background] Alberts DS, Delforge A. Maximizing the delivery of intraperitoneal therapy while minimizing drug toxicity and maintaining quality of life. Semin Oncol. 2006 Dec;33(6 Suppl 12):S8-17. doi: 10.1053/j.seminoncol.2006.11.003. PMID 17223445
- [Background] Armstrong DK, Brady MF. Intraperitoneal therapy for ovarian cancer: a treatment ready for prime time. J Clin Oncol. 2006 Oct 1;24(28):4531-3. doi: 10.1200/JCO.2006.06.7140. No abstract available. PMID 17008690
- [Background] Markman M. Clinical efficacy supporting the role of intraperitoneal drug delivery in the primary chemotherapeutic management of small-volume residual advanced ovarian cancer. Semin Oncol. 2006 Dec;33(6 Suppl 12):S3-7. doi: 10.1053/j.seminoncol.2006.11.002. PMID 17223444
- [Background] Singhal P, Lele S. Intraperitoneal chemotherapy for ovarian cancer: where are we now? J Natl Compr Canc Netw. 2006 Oct;4(9):941-6. doi: 10.6004/jnccn.2006.0077. PMID 17020670
- [Background] Baysal BE, DeLoia JA, Willett-Brozick JE, Goodman MT, Brady MF, Modugno F, Lynch HT, Conley YP, Watson P, Gallion HH. Analysis of CHEK2 gene for ovarian cancer susceptibility. Gynecol Oncol. 2004 Oct;95(1):62-9. doi: 10.1016/j.ygyno.2004.07.015. PMID 15385111
- [Result] Armstrong DK, Bundy BN, Baergen R, et al.: Randomized phase III study of intravenous (IV) paclitaxel and cisplatin versus IV paclitaxel, intraperitoneal (IP) cisplatin and IP paclitaxel in optimal stage III epithelial ovarian cancer (OC): a Gynecologic Oncology Group trial (GOG 172). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-803, 2002.
- [Result] Armstrong DK, Bundy B, Wenzel L, Huang HQ, Baergen R, Lele S, Copeland LJ, Walker JL, Burger RA; Gynecologic Oncology Group. Intraperitoneal cisplatin and paclitaxel in ovarian cancer. N Engl J Med. 2006 Jan 5;354(1):34-43. doi: 10.1056/NEJMoa052985. PMID 16394300
- [Result] DeLoia JA, Krivak T, Darcy KM, et al.: Relationship between the C8092A polymorphisms in ERCC1 and clinical outcome in optimally-resected, stage III epithelial ovarian cancer treated with intraperitoneal or intravenous cisplatin and paclitaxel: a Gynecologic Oncology Group study. [Abstract] American Association for Cancer Research: 98th Annual Meeting, April 14-18, 2007, Los Angeles, CA. A-1674, 2007.
- [Result] Krivak TC, Darcy KM, Tian C, et al.: Relationship between polymorphisms in cordon 118 and C8092A in ERCC1 and clinical outcome in optimally-resected, stage III epithelial ovarian cancer treated with intraperitoneal or intravenous cisplatin and paclitaxel: a Gynecologic Oncology Group study. [Abstract] J Clin Oncol 25 (Suppl 18): A-21050, 733s, 2007.
- [Result] Krivak TC, Darcy KM, Tian C, Armstrong D, Baysal BE, Gallion H, Ambrosone CB, DeLoia JA; Gynecologic Oncology Group Phase III Trial. Relationship between ERCC1 polymorphisms, disease progression, and survival in the Gynecologic Oncology Group Phase III Trial of intraperitoneal versus intravenous cisplatin and paclitaxel for stage III epithelial ovarian cancer. J Clin Oncol. 2008 Jul 20;26(21):3598-606. doi: 10.1200/JCO.2008.16.1323. PMID 18640939
- [Result] Krivak TC, Tian C, Rose GS, Armstrong DK, Maxwell GL. A Gynecologic Oncology Group Study of serum CA-125 levels in patients with stage III optimally debulked ovarian cancer treated with intraperitoneal compared to intravenous chemotherapy: an analysis of patients enrolled in GOG 172. Gynecol Oncol. 2009 Oct;115(1):81-85. doi: 10.1016/j.ygyno.2009.06.021. Epub 2009 Jul 12. PMID 19596139
- [Result] Krivak T, Darcy K, Tian C, et al.: Relationship between polymorphisms in ERCC1 and clinical outcome in optimally resected stage III epithelial ovarian cancer: a Gynecologic Oncology Group study. [Abstract] Society of Gynecologic Oncologists, 2007 Annual Meeting on Women's Cancer, March 3-7, 2007, San Diego, CA. A-146, 2007.
- [Result] Seamon LG, Carlson MJ, Richardson DL, et al.: Improved intraperitoneal chemotherapeutic toxicity profile for ovarian cancer: A modification of the taxane-platinum protocol in GOG-172. [Abstract] J Clin Oncol 26 (Suppl 15): A-5583, 2008.
- [Result] Thrall M, Gallion HH, Kryscio R, Kapali M, Armstrong DK, DeLoia JA. BRCA1 expression in a large series of sporadic ovarian carcinomas: a Gynecologic Oncology Group study. Int J Gynecol Cancer. 2006 Jan-Feb;16 Suppl 1:166-71. doi: 10.1111/j.1525-1438.2006.00504.x. PMID 16515585
- [Result] von Gruenigen VE, Huang HQ, Gil KM, Frasure HE, Armstrong DK, Wenzel LB. The association between quality of life domains and overall survival in ovarian cancer patients during adjuvant chemotherapy: a Gynecologic Oncology Group Study. Gynecol Oncol. 2012 Mar;124(3):379-82. doi: 10.1016/j.ygyno.2011.11.032. Epub 2011 Nov 23. PMID 22119995
- [Result] Walker JL, Armstrong D, Huang H, et al.: Intraperitoneal catheter outcomes on GOG 172: a Gynecologic Oncology Group study in women with optimally debulked stage III ovarian cancer. [Abstract] Int J Gynecol Cancer 14 (Suppl 1): A-062, 19, 2004.
- [Result] Walker JL, Armstrong DK, Huang HQ, Fowler J, Webster K, Burger RA, Clarke-Pearson D. Intraperitoneal catheter outcomes in a phase III trial of intravenous versus intraperitoneal chemotherapy in optimal stage III ovarian and primary peritoneal cancer: a Gynecologic Oncology Group Study. Gynecol Oncol. 2006 Jan;100(1):27-32. doi: 10.1016/j.ygyno.2005.11.013. PMID 16368440
- [Result] Wenzel LB, Huang HQ, Armstrong DK, et al.: Baseline quality of life (QOL) as a predictor of tolerance to intraperitoneal (IP) chemotherapy for advanced epithelial ovarian cancer (EOC): a Gynecologic Oncology Group (GOG) study. [Abstract] J Clin Oncol 24 (Suppl 18): A-5007, 257s, 2006.
- [Result] Wenzel LB, Huang HQ, Armstrong DK, Walker JL, Cella D; Gynecologic Oncology Group. Health-related quality of life during and after intraperitoneal versus intravenous chemotherapy for optimally debulked ovarian cancer: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Feb 1;25(4):437-43. doi: 10.1200/JCO.2006.07.3494. PMID 17264340
- [Result] Wenzel L, Huang HQ, Cella D, Walker JL, Armstrong DK; Gynecologic Oncology Group. Validation of FACT/GOG-AD subscale for ovarian cancer-related abdominal discomfort: a Gynecologic Oncology Group study. Gynecol Oncol. 2008 Jul;110(1):60-4. doi: 10.1016/j.ygyno.2008.02.011. Epub 2008 Apr 21. PMID 18430468